CLINICAL TRIAL: NCT04194788
Title: Prospective Observational Pilot Study on Olfaction Alterations That Occur in Spine Patients After Surgery
Brief Title: Olfaction Changes in Patients Undergoing Spine Surgery
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: TASTEODOR (PI: M Briguglio); L4133 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Orthopedic Disorder of Spine; Smell Disorder
MeSH Terms: conditions — Olfaction Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational prospective study evaluates perioperative olfaction alterations, comprising changes in threshold value, discrimination and identification, which occur in spine patients. The single group is subjected to a preoperative and a postoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* Caucasian race
* Between 50 and 85 years of age
* Candidates to spine surgery
* Acceptance and signing of informed consent

Exclusion Criteria:

* Past or present cancer
* Heart failure
* Kidney failure (III-IV)
* Past or present neuropsychiatric disorders
* Heavy smokers (over/equal 3 cigarettes per day)
* Smell disorders
* Rhinitis
* Allergies to the respiratory system

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spine surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Changes in olfaction threshold | Day before surgery and first day after surgery
  Changes in the olfaction threshold evaluated with a series of solutions having different concentrations of aromas

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided